CLINICAL TRIAL: NCT04866277
Title: Fast-track Referral for Health Interventions During Pregnancy: a Randomized Pragmatic Experimental Study to Reduce Low Birthweight in Portugal
Brief Title: Experimental Study to Reduce Low Birthweight
Acronym: STOP-LBW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Saude Publica da Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CE20140
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Infant, Low Birth Weight
Keywords: Infant, Low Birth Weight; Smoking; Alcohol Drinking; Depression; Physical Abuse; Clinical trial
MeSH Terms: conditions — Smoking; Alcohol Drinking; Depression

STUDY DESIGN:
Intervention Model Description: Parallel superiority pragmatic clinical trial randomized by clusters (Primary Health Care Units)
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, there will be no blinding of pregnant women, health professionals or members of the research team after assignment of the intervention. However, those involved in the outcome assessment and data analysis will be blinded as there will be no identification of the intervention and control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Women who present at least one of the four risk factors - smoking, risk alcohol consumption, risk of depression, physical violence - will be eligible to receive the intervention. The intervention will be the activation of fast-track referral for specialized units and care programs for the four psychosocial and behavioural risk factors under study. All pregnant women referred by the "STOP LBW project" would have access to consultations or other health activities, such as counselling and group meetings, within a maximum of seven days, in reference services available in each metropolitan area. The activation of the fast-track referral will be the responsibility of the doctor/nurse who applies the questionnaires to identify the risk factors. The intervention ends with childbirth, abortion or if the participant decides to abandon the study.
  Interventions: Other: Fast-track referral for reference services
- Standard of care (No Intervention): Women who present at least one of the risk factors - smoking, risk alcohol consumption, risk of depression, physical violence - will receive the standard of care currently existing in each PHCU. The standard of care varies across the various PHCU and may include several approaches: routine screening with care by the antenatal care provider; routine screening with referral to other health professional in the same health unit; and routine screening with referral to other health services, with the time elapsed for consultation depending on the health resources available in each area. In each PHCU, different standards of care may exist for each of the four risk factors.

INTERVENTIONS:
Other: Fast-track referral for reference services — Activation of fast-track referral for specialized units and care programs for the four psychosocial and behavioural risk factors under study.
  Arms: Intervention

SUMMARY:
Introduction: Low birthweight (LBW) is associated with a wide range of short- and long-term consequences and is related to a complex set of maternal psychosocial and behavioural determinants. The objective of this study is to assess the effect of implementing fast-track referral for early intervention on psychosocial and behavioural risk factors - smoking, alcohol consumption, depression and interpersonal violence - on reducing the incidence of LBW.

Methods and analysis: Parallel superiority pragmatic clinical trial randomized by clusters. Primary health care units (PHCU) located in Portugal will be randomized (1:1) to intervention or control groups. Pregnant women over 14 years of age attending these PHCU will be eligible to the study. Risk factors will be assessed through face-to-face interviews. In the intervention group, women who report at least one risk factor will have immediate access to referral services. The comparison group will be the local standard of care for these risk factors. The investigators will use intention-to-treat analyses to compare intervention and control groups. A sample size of 2,832 pregnant women was estimated to detect a 30% reduction in the incidence rate of LBW (primary outcome) between the control and intervention groups. Secondary outcomes are the reduction of preterm births and reduction of risk factors targeted by the intervention.

DETAILED DESCRIPTION:
The investigators will conduct a parallel superiority pragmatic clinical trial randomized by clusters.

The study will be conducted in Primary Health Care Units (PHCU) located in the metropolitan regions of Porto and Lisbon, in Portugal. All 236 PHCU, nested in 13 Primary Care Centres (PCC), will be considered eligible to inclusion (109 PHCU in 7 PCC in Porto; 127 PHCU in 6 PCC in Lisbon).

The investigators will use the PHCU as units of randomization and pregnant/newborn dyads as the unit of analysis. In each of the 13 Primary Care Centres, all PHCU that adhere to the study will be randomized in a 1: 1 ratio for the intervention or control group and will belong to that group until the end of the study. A research team statistician will generate the randomization sequence through Excel Office 365 and implement the random allocation sequence using sequentially numbered, opaque, sealed envelopes.

At each PHCU, all pregnant women, of any gestational age, over the age of 14, who are attending their first prenatal care visit during the study period, that currently reside in Portugal and plan to have a birth in Portugal will be considered eligible and invited to participate in the study.

Health professionals providing prenatal care will be responsible for recruiting pregnant women at their first prenatal visit at the PHCU. Participation in the study is voluntary and non-participation in the study does not affect the routine healthcare provided. The recruitment of participants will last until the planned sample is reached (estimated period of one year).

After being informed of the objectives of the study and giving informed and written consent, pregnant women who agree to participate will answer a face-to-face questionnaire. Data collection will take place in a private environment, that is, in a medical or nursing office, without the presence of other pregnant women, partners or family members, to ensure confidentiality, using an online link.

The electronic questionnaire includes sociodemographic characteristics (date of birth, nationality, marital status, education level, type of work) and risk assessment (smoking, alcohol consume, depression and physical abuse). Considering the particular context of the SARS-CoV-2 pandemic, which can affect intrauterine development of the foetus, the questionnaire also includes information on COVID-19 tests and contact with positive cases. Pregnant women with at least one of the psychosocial or behavioural risk factors will be asked about chronic conditions, medication use, obstetric history, characteristics of the current pregnancy and anthropometry. To assess smoking during pregnancy, the investigators will use a set of questions including pre-pregnancy smoking and smoking during pregnancy (frequency, number of cigarettes per day, gestational month). In women who report smoking during pregnancy, the investigators will assess smoking addiction using the Fagerström nicotine addiction test, validated in Portugal in an academic community of teachers and staff. For alcohol consumption screening, the investigators will use the Alcohol Use Disorders Identification Test - Consumption (AUDIT-C), a scaled-down version of the Alcohol Use Disorders Identification Test (AUDIT), which has a good performance in detecting risky consumption of alcohol during pregnancy. To assess depression, the investigators will use the Portuguese version of the Edinburgh Postpartum Depression Scale (EPDE) with a 9-point cut-off. To assess physical violence against pregnant women the investigators will use the Abuse Assessment Screen (AAS) instrument due to its reliability, validity and easiness of application by clinicians in the context of healthcare provision.

Women who present at least one of the risk factors will be eligible to receive the intervention. The intervention will be the activation of fast-track referral for specialized units and care programs for the four psychosocial and behavioural risk factors under study. All pregnant women referred by the "STOP LBW project" would have access to consultations or other health activities, such as counselling and group meetings, within a maximum of seven days, in reference services available in each metropolitan area. The activation of the fast-track referral will be the responsibility of the doctor/nurse who applies the questionnaires to identify the risk factors. The intervention ends with childbirth, abortion or if the participant decides to abandon the study.

The intervention will have the following process:

i. Any tobacco use during pregnancy = Activation of fast-track referral for smoking cessation consultation in Health Centre Units, Hospitals or other; and/or ii. Risk alcohol consumption (score ≥4 on the test AUDIT-C) = Activation of fast-track referral for consultation in support services for the cessation of alcoholic consumption in Health Centre Units, Hospitals, Division of Intervention in Addictive Behaviours and Dependencies (DICAD), social service or other; and/or iii. Risk of depression (score ≥9 on the EPDE scale) = Activation of fast-track referral for psychology consultation at Health Centre Units, Hospital Psychiatry or other; and/or iv. Physical Violence (affirmative answer to the physical violence question in the AAS) = Activation of the fast-track referral for social service and/or psychological consultation in Health Centre Units, Psychiatry Hospitals, or other.

The control group will be the standard of care currently existing in each PHCU. The standard of care varies across the various PHCU and may include several approaches: routine screening with care by the antenatal care provider; routine screening with referral to other health professional in the same health unit; and routine screening with referral to other health services, with the time elapsed for consultation depending on the health resources available in each area. In each PHCU, different standards of care may exist for each of the four risk factors.

The primary outcome is the incidence of LBW (objective of 30% reduction in the incidence of low birthweight, from 9.0% to 6.5%). The secondary outcomes are: a) the prevalence of each of the four psychosocial and behavioural risk factors (smoking, alcohol consumption, depression and physical violence) at the first prenatal visit and after birth; b) the incidence of preterm births (live births with less than 37 weeks of gestation); and c) the proportion of pregnant women with adherence to care programs targeted at psychosocial and behavioural risk factors and description of the determinants of adherence.

Information on birthweight, gestational age and type of delivery will be obtained from the child health records at the first appointment of the newborn at the PHCU (the moment of the first vaccination will be used whenever possible). The research team will conduct a telephone interview in the first month after birth, using the same screening questionnaire used in the first interview, to assess tobacco and alcohol consumption, the presence of depressive symptoms and exposure to interpersonal violence. The investigators will also measure adherence to care programs aimed at the four risk factors and the determinants of adherence and other strategies used by the pregnant woman to control these risk behaviours.

The sample size was calculated considering the use of bilateral tests, for a significance level of 5% and statistical power of 80%, in order to compare the intervention and control groups in relation to the primary outcome defined in the main objective of the study. It was assumed that the intervention can reduce the incidence of LBW by about 30%, that is, from 9.0% to 6.5%. Estimating an institutional adherence rate of 50%, using an intracluster correlation coefficient of 0.01 (estimated from perinatal health studies in primary health care) 60 and estimating a size variation of 20% in clusters (variation in the number of eligible pregnant women in each PHCU), a sample size of 1,416 participants per intervention / control group was estimated, in a total of 2,832 participants.

Due to the nature of the study, there will be no blinding of pregnant women, health professionals or members of the research team after assignment of the intervention. However, those involved in the outcome assessment and data analysis will be blinded as there will be no identification of the intervention group.

Adherence to the study protocol will be fostered using different strategies including information to pregnant women, project communication through the creation and maintenance of a website, involvement of health professionals during the planning and monitoring phases, and close monitoring of the intervention by the research team. Data collection will be weekly monitored comparing women attended in the first prenatal consultation, women invited to participate and women included in the study. This efforts aim to prevent empty clusters and ensure that the inclusion process of pregnant women is independent of the allocation process.

All questionnaires will be coded using an alphanumeric unique code to ensure confidentiality and anonymity. Clinical and sociodemographic data will be stored in a Limesurvey server from the Institute of Public Health of the University of Porto, to which only two members of the research team will have access (IB and PP). The access to the dataset is private and will only be available by using a specific user account and password. This repository uses digital certificates that guarantee the security of all the communications and traceability. Datasets will be extracted to a SPSS software version 26.0 for analysis and report.

The investigators will conduct an intention-to-treat analysis to compare the results between the intervention and control groups using random effects models that take into account the cluster effect. Pregnant women who have miscarriages; stillbirths; early neonatal deaths without information on birthweight; and pregnant women included in the study who decided to leave the study or who became inaccessible by the research team will be classified as losses to follow-up. The missing data for individual variables will be described and multiple imputation methods used if the missing data is >5%. Characteristics of included women versus losses to follow-up and potential impact on results will be described, with use of statistical techniques, if necessary, to address selection bias. Differences in LBW incidence between the intervention group and the control group clusters will be tested using the chi-square test (χ2) or Fisher's exact test, as appropriate. Adjusted analysis will be conducted to control the effect of potential confounders if maternal characteristics such as age, education, chronic conditions, marital status, type of pregnancy (single or multiple), type of delivery, among others are misbalanced between groups.

A pilot study was conducted from January 8 to June 18, 2020 in ten PHCU including 142 pregnant women (1 refusal, 0.7%). The average gestational age was 19 weeks and 28.2% had at least one of the four risk factors: 14.8% reported smoking during pregnancy, 0.7% had high alcohol consumption, 16.9% had depressive symptoms and 1.4% reported at least one episode of physical abuse during pregnancy.

The investigators had planned to start the clinical trial immediately after the pilot study but it had to be stopped because of the covid-19 pandemic. The study will be resumed in 2021.

Patients and public were not involved in the definition of research questions, outcome measures and design of the study. During the interviews, women will be asked about the burden of the intervention and their acceptance.The investigators intend to involve patients and the public in the plan to disseminate the study results.

All women who agree to participate will sign a written and informed consent. Participants can refuse to participate in the study or withdraw their consent at any time. Refusal or abandonment does not affect the right to receive medical treatment or medical assistance, now or in the future. There is no reason to believe that the intervention will harm the participants. However, all cases of miscarriage, stillbirths, neonatal death, birth defects or maternal death will be recorded. Any potential damage resulting from the investigation will lead to the immediate suspension of part or all of it. The data will be stored electronically on a secure server of the Public Health Institute of the University of Porto (ISPUP), with access only by the research team. All information in the database will be anonymized, using a unique identifier. The key to link the database records and the identification of the participants will be kept by the health professionals of the PHCU.

The results will be disseminated to all health professionals and health service managers in Portugal through meetings and reports. The results will also be made available to pregnant women and the general population through the study website and the press. The main results will be published in scientific journals.

ELIGIBILITY:
Health units:

Inclusion Criteria:

Primary Health Care Units (PHCU) located in the metropolitan regions of Porto and Lisbon, Portugal

Women:

Inclusion criteria: All pregnant women, of any gestational age, over the age of 14, who are attending their first prenatal care visit during the study period, that currently reside in Portugal and plan to have a birth in Portugal.

Exclusion criteria: Pregnant women unable to answer the questionnaire in Portuguese (language barrier, deafness concomitant with blindness, etc.) and/or unable to provide informed consent at the time of recruitment.

Ages: 14 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2832 (Estimated)
Dates: Start 2021-05-02 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Low birthweight | At birth
  Incidence of live births with birthweight < 2500g

SECONDARY OUTCOMES:
Preterm birth | At birth
  Incidence of live births with less than 37 weeks of gestation
Prevalence of risk factors | First prenatal visit and one month after birth
  Prevalence of each of the four psychosocial and behavioural risk factors (smoking, alcohol consumption, depression and physical violence) at the first prenatal visit and after birth
Adherence to care services | One month after birth
  Proportion of pregnant women with risk factors with adherence to care programs targeted at psychosocial and behavioural risk factors and description of the determinants of adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Henrique Barros, Phd, Study Director — Instituto de Saude Publica da Universidade do Porto

IPD SHARING:
Plan to Share IPD: Yes
The protocol of the study will be published in an open access scientific journal. The dataset will be published in a data repository.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Barros H, Baia I, Monjardino T, Pimenta P, Alfredo A, Sorokina A, Domingues R. Fast-track referral for health interventions during pregnancy: study protocol of a randomised pragmatic experimental study to reduce low birth weight in Portugal (STOP LBW). BMJ Open. 2022 Mar 15;12(3):e052964. doi: 10.1136/bmjopen-2021-052964. PMID 35292492